CLINICAL TRIAL: NCT03747081
Title: Comparing Treatment Outcomes in CVT Patients Who Treated With Warfarin and Rivaroxaban in Isfahan, Iran
Brief Title: Efficacy Comparison of Warfarin Versus Rivaroxaban CVT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Saadatnia, Professor Mohammad Saadatnia, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Isfahan Stroke Unit
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Cerebral Venous Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivoroxaban (Experimental): Patients would be administered Enoxaparine (60 mg/SC/BID)in first day, after dicontinuing Enoxaparin in second day, Rivoroxaban 20 mg per day will use. .it would be given once a day.The total duration of Rivoroxaban would be 3 months.
  Interventions: Drug: Rivaroxaban
- warfarin (Active Comparator): Patients would be administered Warfarin with overlap of Enoxaparine utill INR adjust to 2-3 then enoxaparine will disconstinue.it would be given once a day.The total duration of Warfarin would be 3 months
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban will administrate to patient with CVT. In first day, enoxaparin is injected to patients and the next day, patients will receive Rivaroxaban and enoxaparin discontinue. Then, patients receive Rivaroxaban for 3 months daily.
  Other Names: Xarelto
  Arms: Rivoroxaban
Drug: Warfarin — Warfarin as a antocoagolant drug will administrate to patient with CVT. In first day, Warfarin plus enoxaparin until adjusting INR index to 2-3. Then, patients receive warfarin for 3 months daily.
  Other Names: Coumadin
  Arms: warfarin

SUMMARY:
With regard to Cerebral Venous Thrombosis (CVT) importance as a life threatening disease, specific care is necessary, Known anti-coagulants have limitations.Vitamin K antagonists such as Warfarin, require laboratory monitoring and exact administration starting and maintenance dose. although Rivaroxaban(selective and direct Xa factor antagonist ) has no monitoring and no drug interaction. This study aim to focus on efficacy of Warfarin versus Rivaroxaban.

ELIGIBILITY:
IInclusion Criteria:

* Patients of both gender
* Age 18 years and higher
* proven CVT on neuro imaging ( MRI-MRV)

Exclusion Criteria:

* Patients suffering from renal failure(GFR<30) Patients
* Patients with contraindications for oral anticoagulation
* Patient who having pregnancy
* Uncooperative patient for completing the course of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 3 months
  based on disability grade(0-6). 0 indicate patients have no disability and the worst score is 6.

SECONDARY OUTCOMES:
hemorrhagic rate | 3 months
  based on repeat MRI
Stroke | 3 months
  based on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Saadatnia, Prof, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Alzahra University Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957